CLINICAL TRIAL: NCT04730440
Title: Rehabilitation of Facial Emotion Recognition in Alzheimer's Disease and Study of the Consequences on Gaze Strategy, Behavior Disorders and Family Caregivers' Burden
Brief Title: Rehabilitation of Facial Emotion Recognition in Alzheimer's Disease
Acronym: EYE-TAR(MA)
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Princesse Grace (Other)
Collaborators: Association de Recherche Bibliographique pour les Neurosciences (Other); Universite Cote d'Azur (Other)
Responsible Party: Sponsor
Other Study IDs: 19-02
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Alzheimer Dementia; Family Caregivers
Keywords: Video-oculography; Eye-Tracking; Gaze strategies; Oculomotor behaviors; Training of Affect Recognition; Emotion recognition; Facial emotion recognition; Theory of Mind (ToM); Behavioral disorders; Caregiver's burden; Alzheimer's Dementia
MeSH Terms: conditions — Alzheimer Disease; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AD-TAR: AD subjects who take part to Facial Emotion Recognition rehabilitation (TAR)
  Interventions: Other: AD-TAR
- AD-Cognitive Stimulation: AD subjects who take part to cognitive stimulation session (12 sessions during 4 weeks)
  Interventions: Other: AD-Cognitive Stimulation

INTERVENTIONS:
Other: AD-TAR — Intervention description: 12 sessions in groups of 4 subject, over 6 weeks (2 sessions per week), using a rehabilitation program named Training of Affect Recognition (TAR).
  Groups: AD-TAR
Other: AD-Cognitive Stimulation — Intervention description: 12 sessions in groups of 4 subject, over 6 weeks (2 sessions per week), using classic cognitive stimulation workshops.
  Groups: AD-Cognitive Stimulation

SUMMARY:
This study aims to evaluate impacts of an emotion recognition rehabilitation program, named Training of Affect Recognition, on social cognition abilities in Alzheimer's disease (AD). In addition, we hypothesis that the effect of this rehabilitation will also evolve gaze strategies, behavioral disorders, and the caregiver's burden.

DETAILED DESCRIPTION:
It is commonly admitted that social cognition impairment, like deficit in facial emotion recognition or misinterpretation of others' intentions (Theory of Mind), are associated with social behavior disorders.

This kind of disorders are observed in Fronto-Temporal Dementia, Alzheimer's Dementia (AD) and Parkinson's Disease, with severe deficits in FTD and lighter deficits in AD and PD. One explanation is that patients apply inappropriate visual exploration strategies to decode emotions and intentions of others.

Our study aims to evaluate impacts of an emotion recognition rehabilitation program, named Training of Affect Recognition, on social cognition abilities (facial emotion recognition (FER) and theory of mind (ToM)) in Alzheimer's disease (AD). In addition, we hypothesis that the effect of this rehabilitation will also evolve gaze strategies, behavioral disorders, and the caregiver's burden.

ELIGIBILITY:
Inclusion Criteria:

* AD diagnosed according to l'IWG-2 (Dubois & al. 2014) criteria,
* Mini-Mental State (MMS-E) ≥15
* Subject accompanied by a family caregiver and whose participation in a cognitive stimulation workshop was recommended in Memory Centre of the RAINIER Centre (Princesses Grace Hospital - Monaco)
* Written informed consent signed by patient and family caregiver.

Exclusion Criteria:

* General anaesthesia within 3 months.
* Ophthalmological or neurological problems preventing a video-oculography examination.
* Oculomotor disorders such as "fixation disorders" or "ocular tracking disorders".
* Cognitive disorders of the type: visual agnosia, visuo-spatial disorder, visuo-perceptual disorder or aphasia.
* History of bipolar disorder or schizophrenia
* History of alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with an Alzheimer's disease and with a Mini-Mental State score ≥15
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
Facial emotion recognition (FER) performances | Baseline; Week 6; 1 month post intervention
  Change from Baseline and Comparison of FER performance between AD-TAR group and AD-Cognitive Stimulation group.
  Evaluation criteria: Scores to Ekman Faces task (1976) and time to answer. FER was assessed using pictures from the Ekman Faces task (1976), to test the recognition of the six facial basic emotions and neutral faces. There were four pictures per emotion, for a total of 28. For each picture, participants were asked to select one of the seven labels (anger, disgust, fear, sadness, happiness, surprise and neutral), with a maximum of 8 seconds of response time per picture.
Affective ToM performances | Baseline; Week 6; 1 month post intervention
  Change from Baseline and Comparison of Affective ToM performance between AD-TAR group and AD-Cognitive Stimulation group.
  Evaluation criteria: Scores to the " Reading the Mind in the Eyes " test (Baron-Cohen 2001). 36 black-and-white photographs of the eye area of faces. Subjets are asked to choose which word, among four options, best described what the character in the photograph was thinking or feeling. For this task, four scores were obtained: a total score (/36) and three emotional valence sub-scores: positive (/8), neutral (/16) and negative (/12).

SECONDARY OUTCOMES:
Eye gaze strategies during Facial emotion recognition (FER) | Baseline; Week 6; 1 month post intervention
  Change from Baseline and Comparison of gaze patterns between AD-TAR group and AD-Cognitive Stimulation group, during Facial emotion recognition tasks.
  Evaluation criteria: Eye movements (number and duration of fixations on areas of interest) recorded with an eye-tracking device. FER was assessed using some pictures from the Ekman Faces task (1976).
Behavioral disorders | Baseline; Week 6; 1 month post intervention
  Change from Baseline and Comparison between AD-TAR group and AD-Cognitive Stimulation group, Evaluation criteria: Neuropsychiatric Inventory (NPI), a scale that includes ten behavioral items (delusions, hallucinations, agitation, depression, anxiety, euphoria, apathy, disinhibition, irritability and aberrant motor behaviors) and two neurovegetative symptoms (sleep and appetite disorders). The evaluation was based on an interview with patients' primary caregivers. Both the frequency (/5) and the severity (/3) of each behavior were determined and a score was calculated by multiplying the frequency and the severity of each behavior observed during the last month.
The Family caregiver's burden | Baseline; Week 6; 1 month post intervention
  Change from Baseline and Comparison between AD-TAR group and AD-Cognitive Stimulation group, Evaluation criteria: The burden of the family caregiver was measured with the Zarit scale (completed by the caregiver). Composed of 22 questions on the physical, emotional and financial load felt. Total score /88.
Global cognitive performance | Baseline; Week 6; 1 month post intervention
  Change from Baseline and Comparison between AD-TAR group and AD-Cognitive Stimulation group, Evaluation criteria: MMSE (MINI MENTAL STATE EXAMINATION). 30-question general cognitive function assessment. The maximum score is 30.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Remédiation de la reconnaissance des émotions faciales dans la maladie d'Alzheimer et effets sur les stratégies d'observation, les troubles du comportement et le fardeau de l'aidant — https://doi.org/10.1016/j.npg.2020.08.003